CLINICAL TRIAL: NCT00949676
Title: DECIDE-HF - Heart Rate Variability in Heart Failure Patients
Brief Title: DECIDE-HF: Heart Rate Variability in Heart Failure Patients
Acronym: DECIDE-HF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Other Study IDs: DECIDE-HF
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Systolic Heart Failure
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure

SUMMARY:
The purpose of this study is to determine whether heart rate variability-like parameters are related to changes in the disease status of a subject that suffers from a disease that decreases the pumping function of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated the study-specific informed consent form
* Subject is 18 years of age or older
* Subject is expected to remain available for follow-ups
* Subject is able and willing to comply with the protocol requirements
* Subject has predominant Normal Sinus Rhythm
* Subject has systolic Heart Failure and is at the moment of enrollment in NYHA class II or III and has an ejection fraction of less then 40%
* Subject has had a HF-related hospitalization in the past 12 months

Exclusion Criteria:

* Subject needs permanent atrial pacing (> 10%)
* Subject has intermittent 2nd or intermittent 3rd degree block
* Subject has persistent or permanent AF
* Subject has Long QT syndrome, Brugada syndrome, Jervell and Lange- Nielsen syndrome, Romano-Ward syndrome, Andersen-Tawil syndrome or Timothy's syndrome
* Subject has had recent (<2 months) acute coronary syndrome
* Subject has had recent (<2 months) revascularization
* Subject has a pending cardiac transplant or revascularization
* Subject has severe stenotic valvular heart disease
* Subject has severe pulmonary (forced expiratory volume in 1 s < 1 L) hepatic or renal (plasma creatinine > 0.2 mmol/L) disease
* Subject is participating in another study that may affect the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systolic Heart Failure Patients with NYHA class II or III and a ventricular ejection fraction of less then 40%.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
HF diagnostic | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: DECIDE HF Team, Study Chair — Medtronic BRC
Locations (5):
- Antwerp, Belgium
- Germany (3):
  - Kiel
  - Munich
  - Tübingen
- Leeds, United Kingdom